CLINICAL TRIAL: NCT03800849
Title: Mechanical Ventilation Practices and 28-day Patient Mortality in Uganda's Intensive Care Units: A Prospective Cohort Study
Brief Title: Mechanical Ventilation Practices in Uganda's Intensive Care Units
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Other Study IDs: Ventilation
Record Dates: First submitted 2018-09-11; First posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2018-09

CONDITIONS: Mechanically Ventilated Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective cohort study carried out in four ICUs in Uganda. All patients, 18 years and above initiated on mechanical ventilation will be recruited. Patients' data will be collected from the files and charts at initiation of mechanical ventilation. Patients will then be followed up for death / discharge within 28 days in ICU.

DETAILED DESCRIPTION:
Background: The need for mechanical ventilation is one of the commonest indication for admission to the ICU. Despite the clear benefits of mechanical ventilation, it may be detrimental to the patient if poorly carried out. This has led to a renewed impetus in employing lung protective ventilation strategies, Ventilator Associated Events (VAE) prevention strategies, and safe and appropriate weaning methods to reduce mortality among mechanically ventilated patients. However, there is paucity of data regarding these practices in low-income settings.

Objective: To describe the mechanical ventilation practices, mortality rate and associated factors among mechanically ventilated patients in Uganda's intensive care units.

Methodology: A prospective cohort study carried out in four ICUs in Uganda. All patients, 18 years and above initiated on mechanical ventilation will be recruited. Patients' data will be collected from the files and charts at initiation of mechanical ventilation. Patients will then be followed up for death / discharge within 28 days in ICU.

Data analysis: The primary outcome is all-cause mortality during ICU stay. Data will be summarised into means and standard deviations, medians and interquartile ranges and presented in tables, charts, cross-tabulations and graphs. Univariate and multivariate logistic regression will be used to determine factors associated with mortality.

Utility of results: The results from this study will be disseminated to the Ministry of Health and Makerere University in order to plan, standardise and form guidelines regarding mechanical ventilation practices in ICUs in Uganda.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients 18 years and above, initiated on mechanical ventilation, admitted into study ICU during the study period

Exclusion Criteria:

* Patients ventilated in another ICU for more than 24 hours and transferred to study ICUs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated Adult patients in four selected ICUs during the study period who meet the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 214 (Estimated)
Dates: Start 2018-08-14 (Actual); Primary Completion 2019-03-14 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
28 day ICU mortality of mechanically ventilated patients | 7 months
  Patients will be followed up either to discharge or death in ICU to a maximum of 28 days

SECONDARY OUTCOMES:
Duration of mechanical ventilation, ventilatory settings used, use of complementary ICU interventions | 7 months
  At discharge, death or at the end of 28 days, the duration of mechanical ventilation, ventilatory settings used and complementary interventions will be described.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Kyamummi, MBChB, Principal Investigator — Makerere University, Kampala
Locations (1):
- Mulago hospital, Kampala, Uganda